CLINICAL TRIAL: NCT00380445
Title: Effect of Vildagliptin on Adipose Tissue and Skeletal Muscle Metabolism in Obese Patients With Type 2 Diabetes
Brief Title: Effect of Vildagliptin on Fat and Muscle Metabolism in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2379
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Vildagliptin, Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin

SUMMARY:
Please note this study is not being conducted in the United States. The purpose of this study is to test the hypothesis that acute DPP-4 inhibition with vildagliptin improves fat and muscle metabolism in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to complete a 3-week wash-out of current anti-diabetic medication
* Cannot take any medications which may alter gastric motility except for cardiac medication at a stable dose
* Must discontinue beta-blockers and lipid lowering drugs
* Blood glucose criteria must be met
* BMI in the range 30-35

Exclusion Criteria:

* History of type 1 diabetes, diabetes resulting from pancreatic injury, or secondary forms of diabetes
* Need for insulin within 3 months or patients on thiazolidinediones
* Patients taking a sulfonylurea or metformin who cannot safely discontinue medication for the duration of the study
* Significant concomitant disease or complications of diabetes
* Patients with any history of gastrointestinal surgery or positive gastrointestinal symptons
* High tryglycerides as defined by the protocol
* Smokers who cannot abstain from smoking during the treatment periods

Ages: 30 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To explore whether vildagliptin augments insulin mediated inhibition of adipose tissue lipid mobilization following a mixed meal in patients with type 2 diabetes

SECONDARY OUTCOMES:
To measure the effects of vildagliptin on tissue carbohydrate metabolism (skeletal muscle)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Novartis Investigative Site, Investigative Centers, Germany

REFERENCES:
- [Result] Boschmann M, Engeli S, Dobberstein K, Budziarek P, Strauss A, Boehnke J, Sweep FC, Luft FC, He Y, Foley JE, Jordan J. Dipeptidyl-peptidase-IV inhibition augments postprandial lipid mobilization and oxidation in type 2 diabetic patients. J Clin Endocrinol Metab. 2009 Mar;94(3):846-52. doi: 10.1210/jc.2008-1400. Epub 2008 Dec 16. PMID 19088168